CLINICAL TRIAL: NCT01392742
Title: Prospective Observational Study on Predictors of Early On-treatment Response and Sustained Virological Response in HCV-infected Patients Receiving Peginterferon Alfa-2a Plus Ribavirin
Brief Title: An Observational Study on Predictive Factors of Response in Patients With Chronic Hepatitis C Treated With Pegasys (Peginterferon Alfa-2a) and Ribavirin
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25670
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate predictors of early on-treatment response and sustained virological response in patients with chronic hepatitis C receiving Pegasys (peginterferon alfa-2a) and ribavirin. Data will be collected from patients on treatment (24 or 48 weeks) and 24 weeks after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Serologically confirmed chronic hepatitis C (all genotypes)
* Treatment with Pegasys and ribavirin according to the current standard of care and in line with current summaries of product characteristics (SPCs)/local labelling

Exclusion Criteria:

* Coinfection with HIV and/or hepatitis B
* Contraindications according to the SPC for Pegasys/ribavirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis C treated with Pegasys and ribavirin
Sampling Method: Probability Sample
Enrollment: 443 (Actual)
Dates: Start 2011-05-31 (Actual); Primary Completion 2014-07-31 (Actual); Study Completion 2014-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- Bulgaria (9):
  - Mhat - Pleven; Clinic of Gastroenterology, Pleven
  - Umhat St. Georgi; Clinical of Gastroenterology, Plovdiv
  - MHAT Tokuda Hospital Sofia; Department of Gastroenterology at Clinic of Internal Deseases, Sofia
  - UMHAT Alexandrovska EAD; Gastroenterology, Sofia
  - Mhat Queenjoanna; Clinic of Gastroenterology, Sofia
  - Military Medical Academy; Gastroenterology, Sofia
  - Mhat St. Ivan Rilski; Clinic of Gastroenterology, Sofia
  - Mhat St. Zagora; Clinical of Gastroenterology, Stara Zagora
  - Mhat Sveta Marina; Clinic of Gastroenterology, Varna

RESULTS

PARTICIPANT FLOW:
Groups:
- Hepatitis C Virus (HCV) Infected Participants: Participants who were infected by HCV and receiving pegylated interferon alfa-2a (PEG-IFN alfa-2a) 180 micrograms per week (µg/week) subcutaneously, plus ribavirin tablets 1000 milligrams (mg) (those weighing less than [<] 75 kilograms [kg]) or 1200 mg (those weighing greater than [>] 75 kg) orally; were observed for approximately up to 24 weeks after end of treatment (EOT). Dose change was as per investigators' discretion.
Period: Overall Study
Arm/Group | Hepatitis C Virus (HCV) Infected Participants
Started | 443
Completed | 242
Not Completed | 201
Not completed — Premature study termination | 42
Not completed — Failure to return | 35
Not completed — No treatment/no cooperation/withdrew | 12
Not completed — Lost to Follow-up | 34
Not completed — Insufficient therapeutic response (ITR) | 30
Not completed — ITR and Protocol deviation | 1
Not completed — Adverse event/intercurrent illness | 17
Not completed — Protocol Violation | 14
Not completed — Other | 3
Not completed — Missing information | 13

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all screened participants.
Groups:
- HCV Infected Participants: Participants who were infected by HCV and receiving PEG-IFN alfa-2a 180 µg/week subcutaneously, plus ribavirin tablets 1000 mg (those weighing <75 kg) or 1200 mg (those weighing > 75 kg) orally; were observed for approximately up to 24 weeks after EOT. Dose change was as per investigators' discretion.
Arm/Group | HCV Infected Participants
Number analyzed (Participants) | 443
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.61 (12.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182
  Male | 261

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virological Response (SVR)
Description: SVR was defined as undetectable Hepatitis C Virus Ribonucleic Acid (HCV RNA) 24 weeks after completion of the actual treatment period (a single last undetectable HCV RNA Polymerase Chain Reaction [PCR] measured greater than or equal to >=140 days post-treatment).
Time Frame: 24 weeks after End of treatment (EOT) (up to Week 96)
Population: Per Protocol (PP) population included all participants without any protocol violation.
Measure: Number; unit: percentage of participants
Arm/Group | HCV Infected Participants
Number analyzed (Participants) | 331
percentage of participants | 38.7

2. Primary Outcome: Percentage of Participants With Relapse
Description: Relapse was define as аn undetectable HCV RNA during the treatment period, but without such during the follow-up.
Time Frame: Up to 24 weeks after EOT (up to Week 96)
Population: PP population.
Measure: Number; unit: percentage of participants
Arm/Group | HCV Infected Participants
Number analyzed (Participants) | 331
percentage of participants | 8.2

3. Primary Outcome: Percentage of Participants Who Were Non-Responders
Description: Non-responders were those participants who had not reached аn undetectable HCV RNA during the treatment period.
Time Frame: Up to 24 weeks after EOT (up to Week 96)
Population: PP population.
Measure: Number; unit: percentage of participants
Arm/Group | HCV Infected Participants
Number analyzed (Participants) | 331
percentage of participants | 25.1

4. Secondary Outcome: Percentage of Participants With Positive Predictive Value on SVR at Week 4
Description: Predictive value determined the relationship of the virological response at specified time to the total response. Positive predicted value= number of true positives/(number of true positives+ number of false positives). SVR was defined as undetectable HCV RNA 24 weeks after end of treatment. Percentage of participants who showed positive predictive value in treatment naive and those who failed previous treatment with interferon were reported.
Time Frame: Week 4
Population: PP population. Here "number of participants analyzed" included participants who were evaluable for this outcome measure and "n" signified evaluable participants for specific group.
Measure: Number; unit: percentage of participants
Arm/Group | HCV Infected Participants
Number analyzed (Participants) | 187
percentage of participants
  Treatment naive(n=182) | 64.8
  Failed previous treatment(n=5) | 20.0

5. Secondary Outcome: Percentage of Participants With Positive Predictive Value on SVR at Week 12
Description: Predictive value determined the relationship of the virological response at specified time to the total response. Positive predicted value= number of true positives/( number of true positives+ number of false positives). SVR was defined as undetectable HCV RNA 24 weeks after end of treatment. Percentage of participants who showed positive predictive value in treatment naive and those who failed previous treatment with interferon were reported.
Time Frame: Week 12
Population: PP population. Here "number of participants analyzed" included participants evaluable for the outcome measure and "n" signified evaluable participants for specific group.
Measure: Number; unit: percentage of participants
Arm/Group | HCV Infected Participants
Number analyzed (Participants) | 186
percentage of participants
  Treatment naive(n=182) | 69.8
  Failed previous treatment(n=4) | 25.0

6. Secondary Outcome: Correlation of SVR With Rapid Virological Response (RVR)
Description: Correlation of SVR with RVR was based on 3 symmetric measures; Kendall's tau-b, Kendall's tau-c and Gamma. SVR was defined as undetectable HCV RNA 24 weeks after end of treatment. RVR was defined as having undetectable HCV RNA 4 weeks after start of treatment.
Time Frame: Up to 24 weeks after EOT (up to Week 96)
Population: PP population. Here "number of participants analyzed" included participants who were evaluable for this outcome measure.
Measure: Number; unit: correlation coefficient
Arm/Group | HCV Infected Participants
Number analyzed (Participants) | 238
correlation coefficient
  Kendall's tau-b | 0.378
  Kendall's tau-c | 0.310
  Gamma | 0.782

7. Secondary Outcome: Correlation of SVR With Early Virological Response (EVR)
Description: Correlation of SVR with EVR was based on 3 symmetric measures; Kendall's tau-b, Kendall's tau-c and Gamma. SVR was defined as undetectable HCV RNA 24 weeks after end of treatment. EVR was defined as having undetectable HCV RNA 12 weeks after start of treatment.
Time Frame: Up to 24 weeks after EOT (up to Week 96)
Population: PP population. Here "number of participants analyzed" included participants who were evaluable for this outcome measure.
Measure: Number; unit: correlation coefficient
Arm/Group | HCV Infected Participants
Number analyzed (Participants) | 238
correlation coefficient
  Kendall's tau-b | 0.570
  Kendall's tau-c | 0.470
  Gamma | 1.000

8. Secondary Outcome: Predictive Power Values of Host-, Virus- and Treatment-related Factors and Virological Response
Description: Predictive value determined the relationship of host factors to virological response. Host factors included; RVR (EVR for Week 12), gender, liver fibrosis, HCV genotype, height and treatment duration for Week 4 after EOT excluding HCV genotype at Week 12 EOT. RVR was defined as having undetectable HCV RNA 4 weeks after start of treatment and EVR was defined as having undetectable HCV RNA 12 weeks after start of treatment.
Time Frame: Week 4 and 12
Population: PP population. Here "number of participants analyzed" included participants who were evaluable for this outcome measure
Measure: Number; unit: predictive value
Arm/Group | HCV Infected Participants
Number analyzed (Participants) | 238
predictive value
  Week 4: RVR | 2.540
  Week 4: gender | 1.390
  Week 4: liver fibrosis | 7.030
  Week 4: HCV genotype | 2.320
  Week 4: height | -0.091
  Week 4: treatment duration | 0.020
  Week 12: EVR | 5.860
  Week 12: gender | 1.291
  Week 12: liver fibrosis | 4.774
  Week 12: height | -0.071
  Week 12: treatment duration | 0.006
Statistical Analysis 1: Comparison: HCV Infected Participants; Binary logistic regression for RVR at Week 4; Test type: Superiority or Other; p = 0.000, Regression, Logistic
Statistical Analysis 2: Comparison: HCV Infected Participants; Binary logistic regression for gender at Week 4; Test type: Superiority or Other; p = 0.018, Regression, Linear
Statistical Analysis 3: Comparison: HCV Infected Participants; Binary logistic regression for liver fibrosis at Week 4; Test type: Superiority or Other; p = 0.062, Regression, Logistic
Statistical Analysis 4: Comparison: HCV Infected Participants; Binary logistic regression for HCV genotype at Week 4; Test type: Superiority or Other; p = 0.050, Regression, Logistic
Statistical Analysis 5: Comparison: HCV Infected Participants; Binary logistic regression for height at Week 4; Test type: Superiority or Other; p = 0.001, Regression, Logistic
Statistical Analysis 6: Comparison: HCV Infected Participants; Binary logistic regression for treatment duration at Week 4; Test type: Superiority or Other; p = 0.001, Regression, Logistic
Statistical Analysis 7: Comparison: HCV Infected Participants; Binary logistic regression for EVR at Week 12; Test type: Superiority or Other; p = 0.037, Regression, Logistic
Statistical Analysis 8: Comparison: HCV Infected Participants; Binary logistic regression for gender at Week 12; Test type: Superiority or Other; p = 0.018, Regression, Logistic
Statistical Analysis 9: Comparison: HCV Infected Participants; Binary logistic regression for liver fibrosis at Week 12; Test type: Superiority or Other; p = 0.092, Regression, Logistic
Statistical Analysis 10: Comparison: HCV Infected Participants; Binary logistic regression for height at Week 12; Test type: Superiority or Other; p = 0.001, Regression, Logistic
Statistical Analysis 11: Comparison: HCV Infected Participants; Binary logistic regression for treatment duration at Week 12; Test type: Superiority or Other; p = 0.042, Regression, Logistic

9. Secondary Outcome: Duration of Treatment in Participants With SVR by HCV Genotype
Description: SVR was defined as undetectable HCV RNA 24 weeks after end of treatment.
Time Frame: Up to Week 72
Population: PP population. Here "number of participants analyzed" included participants evaluable for the outcome measure and "n" signified evaluable participants for specific HCV genotype.
Measure: Mean (Full Range); unit: days
Arm/Group | HCV Infected Participants
Number analyzed (Participants) | 128
days
  HCV genotype 1(n=111) | 329.95 [116.00 to 365.00]
  HCV genotype 3(n=16) | 173.25 [140.00 to 337.00]
  HCV genotype 4(n=1) | 335.00 [335.00 to 335.00]

10. Secondary Outcome: Cumulative PEG-IFN Alfa-2a Dose in Participants With SVR by HCV Genotype
Description: SVR was defined as undetectable HCV RNA 24 weeks after end of treatment.
Time Frame: Up to Week 72
Population: as for outcome 9
Measure: Mean (Full Range); unit: µg
Arm/Group | HCV Infected Participants
Number analyzed (Participants) | 128
µg
  HCV genotype 1(n=111) | 24701.70 [6711.43 to 28157.14]
  HCV genotype 3(n=16) | 13030.71 [10800.00 to 25997.14]
  HCV genotype 4(n=1) | 25842.86 [25842.86 to 25842.86]

11. Secondary Outcome: Cumulative Ribavirin Dose in Participants With SVR by HCV Genotype
Description: SVR was defined as undetectable HCV RNA 24 weeks after end of treatment.
Time Frame: Up to Week 72
Population: as for outcome 9
Measure: Mean (Full Range); unit: mg
Arm/Group | HCV Infected Participants
Number analyzed (Participants) | 128
mg
  HCV genotype 1(n=111) | 1062607 [348000.00 to 1314000]
  HCV genotype 3(n=16) | 538812.50 [100800.00 to 1011000]
  HCV genotype 4(n=1) | 1005000 [1005000 to 1005000]

12. Secondary Outcome: Percentage of Participants With Virological Response
Description: The Virological response at the end of treatment was defined as the percentage of participants with undetectable HCV RNA, HCV test (based on a single last undetectable HCV RNA PCR falling in the 4 weeks' time window at end of treatment), is basically the sum of participants with SVR and with relapse.
Time Frame: 4 weeks after EOT (up to Week 76)
Population: PP population.
Measure: Number; unit: percentage of participants
Arm/Group | HCV Infected Participants
Number analyzed (Participants) | 331
percentage of participants | 46.8

ADVERSE EVENTS:
Time Frame: 24 weeks after EOT (up to Week 96)
Description: Safety population included all participants with any therapy assessment.
Groups:
- HCV Infected Participants: Participants who were infected by HCV and receiving PEG-IFN alfa-2a 180 µg/week subcutaneously, plus ribavirin tablets 1000 mg (those weighing <75 kg) or 1200 mg (those weighing > 75 kg) orally; were observed for approximately 24 weeks. Dose change was as per investigators' discretion.
Arm/Group | HCV Infected Participants
Serious Adverse Events (participants affected / at risk) | 17/440
Other Adverse Events (participants affected / at risk) | 273/440
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HCV Infected Participants (N=440)
Anaemia (Blood and lymphatic system disorders) | 4
Anaemia haemolytic (Blood and lymphatic system disorders) | 1
Astenia (Blood and lymphatic system disorders) | 1
Leucopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Chronic gastritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 2
Drug reaction with eosinophilia and systemic symptoms (Immune system disorders) | 1
Latent tuberculosis (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
Cerebral infarction (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Ischeamic stroke (Nervous system disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Renal abcess (Renal and urinary disorders) | 1
Renal sepsis (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Hypotonia (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HCV Infected Participants (N=440)
Anaemia (Blood and lymphatic system disorders) | 114
Leucopenia (Blood and lymphatic system disorders) | 115
Thrombocytopenia (Blood and lymphatic system disorders) | 111
Fever (General disorders) | 68
Fatigue (General disorders) | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.